CLINICAL TRIAL: NCT02803957
Title: Randomized Trial of the NeoChord™ DS1000™ System Versus Open Surgical Repair
Brief Title: Randomized Trial of the Neochord DS1000 System Versus Open Surgical Repair
Acronym: ReChord
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NeoChord (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NeoChord: PR-610405-100
Record Dates: First submitted 2016-05-09; First posted 2016-06-17 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Mitral Valve Insufficiency
Keywords: Degenerative; Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): Subjects with degenerative mitral valve insufficiency treated with artificial chordae implanted using the NeoChord DS1000
  Interventions: Device: NeoChord DS1000
- Control Group (Active Comparator): Subjects with degenerative mitral valve insufficiency treated with standard surgical mitral valve repair
  Interventions: Device: Surgical Mitral Valve Repair

INTERVENTIONS:
Device: NeoChord DS1000 — Trans-apical, beating heart repair of degenerative mitral valve insufficiency with artificial chordae implanted with the NeoChord DS1000
  Arms: Treatment Group
Device: Surgical Mitral Valve Repair — Surgical repair of degenerative mitral valve insufficiency with cardiopulmonary bypass, and annuloplasty ring and some form of leaflet repair or artificial chordae.
  Arms: Control Group

SUMMARY:
The objective of this trial is to assess the safety and effectiveness of the study device in subjects with degenerative mitral valve disease receiving a mitral valve repair without cardiopulmonary bypass (treatment group) when compared to subjects receiving mitral valve repair using standard surgical techniques with cardiopulmonary bypass (control group).

ELIGIBILITY:
Inclusion Criteria:

* Is a candidate for mitral valve repair with cardiopulmonary bypass
* Has Grade III moderate or Grade IV severe degenerative mitral valve regurgitation
* Primary segmental prolapse of the A2 or P2 segment or prolapse extending to an adjacent segment (P1, P3, A1, A3) who have a single eccentric regurgitant jet on echocardiogram
* Anterior leaflet covers at least 65% of anterior-posterior annular distance or an anterior leaflet that would provide sufficient coaptation after chord placement
* Anatomic and general suitability

Exclusion Criteria:

* Prior mitral valve surgery
* Concomitant cardiac procedures
* Other cardiac procedures within 3 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 585 (Estimated)
Dates: Start 2016-11-03 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects free of Major Adverse Events (MAEs) in the treatment group when compared to subjects in the control group. | Post-operative Day (POD) 30
Proportion of subjects free of Grade II, III or IV mitral regurgitation, mitral valve replacement or mitral valve reintervention in the treatment group when compared to subjects in the control group. | 1 year

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Sutter Health/Alta Bates Summitt Medical Center, Oakland, California
  - Mercy General Hospital, Sacramento, California
  - Stanford University, Stanford, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Hospital, Orlando, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Franciscan Health, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mount Sinai, Icahn School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Pinnacle Health, Harrisburg, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - St. Thomas, Nashville, Tennessee
  - Baylor - Plano, Plano, Texas
  - Valley Health System | Virginia, Winchester, Virginia

IPD SHARING:
Plan to Share IPD: No